CLINICAL TRIAL: NCT00193830
Title: High Dose Rate (HDR) Versus Low Dose Rate (LDR) Brachytherapy in Carcinoma Cervix
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tata Memorial Hospital (Other Government)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: TMH/11062/1996/Cx_HDR STUDY
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2007-01

CONDITIONS: Cancer of Cervix; Cervical Cancer; Cancer of the Cervix; Cervix Cancer
Keywords: Cervical Cancer; High Dose Rate (HDR) Brachytherapy; Low Dose Rate (LDR) Brachytherapy; Acute Toxicities; Late Radiation Sequelae
MeSH Terms: conditions — Uterine Cervical Neoplasms; Barakat syndrome

INTERVENTIONS:
Procedure: HIgh Dose Rate Vs Low DOse Rate Brachytherapy

SUMMARY:
Radiation therapy still remains mainstay of treatment for patients with carcinoma cervix in advanced stages. Conventional treatment with radiation therapy includes a combination of external beam radiation therapy and intracavitary treatment. Low dose rate intracavitary brachytherapy treatment is the time-tested modality of brachytherapy with sound radiobiological bases. But high dose rate brachytherapy is a relatively new alternative. In low dose rate brachytherapy the staff receives some radiation while in the high dose rate brachytherapy procedure complete protection to staff can be achieved as the treatment is done with remote afterloading technique. The high dose rate brachytherapy is possible as Out Patient Department procedure. Few clinical trials have proven the feasibility and efficacy of high dose rate brachytherapy in carcinoma of cervix. However, there is no concrete evidence especially in developing countries for the change of practice to HDR brachytherapy. Hence, at Tata Memorial Hospital with an aim to assess the efficacy, feasibility, early and late complications of high dose rate brachytherapy in contrast with low dose rate brachytherapy we propose this study.

DETAILED DESCRIPTION:
Carcinoma cervix is the most common malignancy in Indian women and constitutes approximately 27% of all cancers as recorded in the annual report of Hospital based cancer registry 1991. Carcinoma of cervix forms one of the leading causes for death and disability due to cancers in India.

Nearly 80% of the patients with carcinoma cervix present in advanced stages. Despite the advances in conventional modalities the five-year survival is 26% and 43% for stage IIIB and stage IIB respectively. In developing countries the socio-economic problems, illiteracy, late presentation and irregular follow-up resulting in early locoregional and distant failures further compound the problem.

Radiation therapy still remains the important modality of treatment for patients with carcinoma cervix in advanced stages. Conventional treatment with radiation therapy includes a combination of external beam radiation therapy and intracavitary treatment. Low dose rate intracavitary treatment is the time-tested modality of brachytherapy for carcinoma of cervix having sound radiobiological bases. But high dose rate brachytherapy is a relatively new method. In low dose rate brachytherapy the staff receives some radiation while in the high dose rate brachytherapy procedure complete protection to staff can be achieved as the treatment is done with remote afterloading technique. The high dose rate brachytherapy is possible as OPD procedure. Various clinical trials have proved the feasibility and efficacy of high dose rate brachytherapy for carcinoma of cervix. At Tata Memorial Hospital we advocate a study to assess the efficacy, feasibility, early and late complications of high dose rate brachytherapy in contrast with low dose rate brachytherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven squamous carcinoma of cervix
* Performance index WHO grade 0 or 1
* Patients below 65 years of age
* Normal ECG and CVS
* Normal hematological parameters
* Normal renal and liver function tests

Exclusion Criteria:

* Concomitant disease which may adversely affect the outcome
* Poor nutritional status
* Medical or psychological condition precluding treatment
* Previous treatment

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750
Dates: Start 1996-05; Study Completion 2007-01

PRIMARY OUTCOMES:
To asses the feasibility of high dose rate brachytherapy
To compare the early and late reactions of high dose rate brachytherapy in contrast with low dose rate brachytherapy.
To compare the over-all survival and disease free survival in the two regimens.

CONTACTS AND LOCATIONS:
Overall Officials: Shyamkishore J Shrivastava, MD, DNB (RT), Principal Investigator — Professor & Head, Radiation Oncology, Tata Memorial Hospital
Locations (1):
- Tata Memorial Hospital, Mumbai, Maharashtra, India